CLINICAL TRIAL: NCT00798837
Title: A Dose-escalation Study Using a Maximal Simultaneous Intraprostatic Boost With RapidArc Intensity Modulated Radiotherapy in Intermediate Risk Prostate Cancer
Brief Title: Intraprostatic MAXimal Simultaneous Boost
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Excess risk in rectal bleeding of first 10 patients
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Principal Investigator, James Morris, Dr. James Morris, British Columbia Cancer Agency
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMAX
Record Dates: First submitted 2008-11-24; First posted 2008-11-26 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Prostate Cancer
Keywords: prostate; cancer; IMRT; radiation
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IMAX (Other): There is only one arm in this study.
  Each patient will undergo a course of intensity modulated external beam radiation therapy (IMRT) using RapidArc for optimization and delivery.
  Doses of radiotherapy are as follows:
  * The prescription dose will be 73.7 Gy in 28 fractions.
  * A simultaneous intraprostatic maximal simultaneous boost will be given to as much of the CTV as possible without contravening OAR dose constraints.
  Interventions: Radiation: Intraprostatic maximal simultaneous boost

INTERVENTIONS:
Radiation: Intraprostatic maximal simultaneous boost — Each patient will undergo a course of intensity modulated external beam radiation therapy (IMRT) using RapidArc for optimization and delivery.
  Doses of radiotherapy are as follows:
  * The prescription dose will be 73.7 Gy in 28 fractions
  * A simultaneous intraprostatic boost will be given to as much of the CTV as possible without contravening OAR dose constraints.

SUMMARY:
This trial uses a type of radiotherapy called intensity modulated radiotherapy (IMRT), which is able to deliver the radiation to the prostate while delivering less dose to the surrounding normal organs compared with standard 3D conformal radiotherapy presently used at the BCCA. This trial will use RapidArc IMRT, which is a new way of delivering IMRT, where the radiation dose is delivered in a single rotation of the radiotherapy machine around the patient. This new method of delivering IMRT has been shown to be at least as good as conventional IMRT at delivering the dose, and takes less time to do so.

The aim of this study is to deliver a higher radiation dose to the prostate gland than the standard treatment while not increasing dose to the normal organs. In this way, it is hoped that the likelihood of the cancer coming back will be reduced without causing an increase in side-effects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically proven adenocarcinoma of the prostate.
2. Registration must occur within 26 weeks of biopsy.
3. History and physical examination (including digital rectal examination (DRE)) within 8 weeks prior to registration.
4. Patients must have intermediate risk prostate cancer, as defined by:

   * PSA ≤ 20 ng/ml,
   * Gleason ≤ 7,
   * Stage ≤ T2c, and
   * Do not meet criteria for low-risk prostate cancer (Low-risk = All of: PSA ≤ 10 + Gleason ≤ 6 + stage ≤ T2b)
5. Patients must have the following blood tests within two weeks of registration:

   * Prostate specific antigen (PSA), testosterone (TTT), complete blood count (CBC), electrolytes, creatinine.
   * Patients with values for one or more of these tests (not including PSA) that fall outside the normal range will need to be reviewed by the oncologist to determine their eligibility for this study.
6. Patients must have an estimated life expectancy of at least 10 years.
7. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2.
8. Patients must have no contraindications to high dose pelvic irradiation.
9. Patients must not have received prior radiation therapy to the pelvis.
10. Patients must have no history of inflammatory bowel disease.
11. Patients must not have received prior hormonal therapy or chemotherapy.
12. Patients must not have any hormonal therapy planned as part of the therapeutic intervention.
13. Patients must have no contraindication to MRI scanning.
14. Patients should not have an artificial hip
15. Patients should not have a body mass index (BMI) of > 32. Note: BMI = weight in kg ÷ (height in metres)2

Exclusion Criteria:

1. Subjects that do not meet inclusion criteria.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-12; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Incidence of grade 2-4 gastrointestinal and genitourinary toxicity | No time frame (post-treatment)

SECONDARY OUTCOMES:
Quality of life (EPIC, IPSS and SHIM questionnaires) | Post-treatment; every 6 mos until 5 years - then annual
Percentage of CTV treated to boost dose | Immediately post-treatment
Time-cost analysis compared to external-beam radiotherapy with brachytherapy boost | No time frame
Accuracy of surrogate urethra compared to T2-MRI localization | No time frame
Quantification of dose received by lesions identified by diffusion-weighted and dynamic contrast enhanced MRI | No time frame

CONTACTS AND LOCATIONS:
Overall Officials: William J Morris, MD, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- British Columbia Cancer Agency - Vancouver Centre, Vancouver, British Columbia, Canada